CLINICAL TRIAL: NCT05433077
Title: Real Life Pacthe : Support and Post-therapeutic Rehabilitation for Women in Complete Remission of Breast Cancer in a Thermal Environment
Brief Title: Support and Post-therapeutic Rehabilitation for Women in Complete Remission of Breast Cancer in a Thermal Environment
Acronym: PACTHE-VR
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Collaborators: Conseil National des Etablissements Thermaux (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-A00171-42
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Non-Metastatic Breast Carcinoma; Remission; Quality of Life
Keywords: Non-metastatic Breast cancer; Spa therapy; remission; Quality of life; supportive care; Post-cancer rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The PACThe - Real life project is a post-therapeutic support and rehabilitation for women in complete remission of breast cancer in a thermal environment. It consists of a 3 weeks spa treatment for patients in remission of breast cancer. This stay in spa treatment will be an adapted "post-cancer" support and has the main objective of showing a lasting improvement in the quality of life following the program offered to women following their breast cancer treatments.

The evaluation of the quality of life will be done using the SF-36 self-questionnaire which will be completed by the patients 5 times (inclusion visit, end of the spa stay, 6 months post-cure, 12 months post-cure and 18 months post-cure).

DETAILED DESCRIPTION:
Post-cancer rehabilitation has developed over the past twenty years. Among the support care put in place, there are in particular thermal cures. On the prescription of a doctor, they represent a medical treatment consisting in exploiting the thermal waters in order to help the recovery of patients.

Several studies have been carried out on the subject, in which it has been shown that spa treatments improve physical and emotional well-being, quality of life and also limit the occurrence of treatment-related toxicities.

The PACThe study, conducted in the thermal spas of Châtel-Guyon, Mont-Dore and Vichy and whose promoter was the Center Jean Perrin, showed that thermal cures significantly improved depression, the quality of sleep as well as quality of life of patients in remission from breast cancer. Following these conclusive results, the CNETh and the UNCAM agreed to set up a post-cancer rehabilitation program covered at 50% by social security, in multiple thermal centers in France. At the same time, the CNETh set up the PACThe-real-life study, which would back up this post-cancer program, in order to confirm and verify the reproducibility of the results of the PACThe study at the national level.

The PACThe-real-life study is an observational RIPH 3 type study with longitudinal cohort follow-up during a post-therapeutic support and rehabilitation program in a spa environment. This study plans to recruit patients aged 20 to 75, in remission from breast cancer, and whose treatment has been completed.

The cures contain a complete program of approximately 3 weeks, composed not only of baths, but also of physical activity, aquagymnastics, massage and physiotherapy, as well as dietary and psychological monitoring. All this allowing the physical, social, professional, family and psychological reconstruction of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from breast cancer
* Treated by chemotherapy and/or radiotherapy
* Absence of residual or progressive disease
* Patient whose treatment has ended (except hormone therapy)
* Able to give informed consent to participate in research
* Affiliation to a Social Security scheme

Exclusion Criteria:

* Cancer in progressive or metastatic phase
* Disabled patient
* Serious personality or eating behavior disorders (craving, bulimia, etc.)
* Thinness (BMI < 18.5 kg.m-2)
* Severe to massive obesity (BMI > 35 kg.m-2)
* Refusal to participate
* Contraindication to physical activity (of cardiovascular origin or linked to a pathology of the musculoskeletal system), lymphedema is not a contraindication
* Participation in another clinical study
* Insufficient knowledge or understanding of the French language making it impossible to correctly complete a self-administered quality of life questionnaire or to answer a dietary questionnaire
* The medical contraindications of spa treatment validated by the French Society of Hydrology and Climatology will be applied and are as follows:
* Severe alterations in general condition (evolving infectious state, renal or hepatic insufficiency, cirrhosis, respiratory insufficiency, etc.)
* Severe or acute ulcerative colitis and Crohn's disease
* Severe immunodeficiencies
* Recent phlebitis
* Hypertension

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 75, suffering from breast cancer and having been treated with chemotherapy and/or radiotherapy, currently in complete remission who are going to undergo a spa treatment as part of the post-cancer programme.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life SF-36 | 6 months after inclusion
  Global score of the short-form 36 (SF-36) quality of life questionnaire. The score goes from 0 to 100. Higher is the score, better is the quality of life.

SECONDARY OUTCOMES:
Quality of life SF-36 (Global scores) | up to 18 months
  Global scores of the short-form 36 (SF-36) quality of life questionnaire. The score goes from 0 to 100. Higher is the score, better is the quality of life.
Quality of life SF-36 (Scores of the subscales) | up to 18 months
  Scores of the subscales of the short-form 36 (SF-36) questionnaire. The score goes from 0 to 100. Higher is the score, better is the quality of life.
Quality of life SF-36 by subgroups | 6 months after inclusion
  Global scores of the SF-36 quality of life questionnaire by subgroups (BMI, age, menopausal status, level of education, precariousness (evaluated via the EPICES score)). The score goes from 0 to 100. Higher is the score, better is the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Dr/Pr, Study Director — Centre Jean Perrin
Locations (15):
- France (15):
  - Thermes de Balaruc-les-Bains, Balaruc-les-Bains
  - Thermes de Barbotan, Barbotan-les-Thermes
  - Thermes de Cambo-les-Bains, Cambo-les-Bains
  - Thermes de Capvern-les-Bains, Capvern
  - Thermes de Contrexéville, Contrexéville
  - Bains de Sarrailh, Dax
  - Thermes d'Eugénie-les-Bains, Eugénie-les-Bains
  - Thermes de Gréoux-les-Bains, Gréoux-les-Bains
  - Thermes de La Léchère, La Léchère
  - Thermes de la Roche-Posay, La Roche-Posay
  - Thermes de Luxeuil-les-Bains, Luxeuil-les-Bains
  - Thermes de Molitg-les-Bains, Molitg-les-Bains
  - Thermes de Saint Amand-les-Eaux, Saint-Amand-les-Eaux
  - Thermes de Soucéo, Saint-Paul-lès-Dax
  - Thermes de Saujon, Saujon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwiatkowski F, Mouret-Reynier MA, Duclos M, Leger-Enreille A, Bridon F, Hahn T, Van Praagh-Doreau I, Travade A, Gironde M, Bezy O, Lecadet J, Vasson MP, Jouvency S, Cardinaud S, Roques CF, Bignon YJ. Long term improved quality of life by a 2-week group physical and educational intervention shortly after breast cancer chemotherapy completion. Results of the 'Programme of Accompanying women after breast Cancer treatment completion in Thermal resorts' (PACThe) randomised clinical trial of 251 patients. Eur J Cancer. 2013 May;49(7):1530-8. doi: 10.1016/j.ejca.2012.12.021. Epub 2013 Jan 24. PMID 23352440
- [Background] Mourgues C, Gerbaud L, Leger S, Auclair C, Peyrol F, Blanquet M, Kwiatkowski F, Leger-Enreille A, Bignon YJ. Positive and cost-effectiveness effect of spa therapy on the resumption of occupational and non-occupational activities in women in breast cancer remission: a French multicentre randomised controlled trial. Eur J Oncol Nurs. 2014 Oct;18(5):505-11. doi: 10.1016/j.ejon.2014.04.008. Epub 2014 May 29. PMID 24882370
- [Background] Kwiatkowski F, Mouret-Reynier MA, Duclos M, Bridon F, Hanh T, Van Praagh-Doreau I, Travade A, Vasson MP, Jouvency S, Roques C, Bignon YJ. Long-term improvement of breast cancer survivors' quality of life by a 2-week group physical and educational intervention: 5-year update of the 'PACThe' trial. Br J Cancer. 2017 May 23;116(11):1389-1393. doi: 10.1038/bjc.2017.112. Epub 2017 Apr 20. PMID 28427084
- [Derived] Godiveau M, Passildas J, Thivat E, Casile M, Pinard C, Giro A, Mouret-Reynier MA, Molnar I, Abrial C, Bouvier CE, Bignon YJ, Durando X. Post-therapeutic support and rehabilitation for breast cancer women in complete remission in a thermal resort: study protocol for the PACThe Real-Life conditions observational trial. BMC Cancer. 2025 Jan 29;25(1):174. doi: 10.1186/s12885-025-13524-2. PMID 39881247